CLINICAL TRIAL: NCT03955081
Title: Safety and Performance of the Motorized Spiral Endoscope (PowerSpiral) in Subjects Indicated for Small-bowel Enteroscopy: A PMCF Registry
Brief Title: A Clinical Study With the Medical Device PowerSpiral for Deep Enteroscopy
Acronym: SAMISEN
Status: Completed | Type: Observational
Sponsor: Olympus Europe SE & Co. KG (Industry)
Responsible Party: Sponsor
Other Study IDs: 2018-GI (OEKG) - 01
Record Dates: First submitted 2019-02-01; First posted 2019-05-17 (Actual); Results first posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2020-08

CONDITIONS: Small Bowel Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Deep enteroscopy — A deep enteroscopy conducted with the new medical device PowerSpiral.

SUMMARY:
The objective of the SAMISEN study is to assess the performance and safety of diagnostic and therapeutic procedures with the newly designed Olympus Motorized Spiral Enteroscope (PowerSpiral).

DETAILED DESCRIPTION:
The main objective of this registry is to collect data on the safety and performance of the new motorized PowerSpiral device during Post-market Clinical Follow-up. It is assumed that the new device and its safety profile is non-inferior to preceding generations of balloon assisted enteroscopes.

As clinical performance and efficacy is equally important for the user this study also collects efficacy and handling data of the new device.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Patients with small bowel disease indicated for deep enteroscopy

Exclusion Criteria:

1. Age under 18 years
2. Female and of child-bearing age who is currently pregnant or planning to become pregnant within the study period
3. Any contraindication to standard enteroscopy
4. Concurrent participation in another competing clinical study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with an indication for direct visualization of the small bowel which fulfil all of these inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 302 (Actual)
Dates: Start 2019-09-02 (Actual); Primary Completion 2021-03-23 (Actual); Study Completion 2021-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Torsten Beyna, MD, Principal Investigator — Evangelisches Kranken-haus Düssel-dorf
Locations (10):
- Belgium (2):
  - Cliniques universitaires Saint-Luc ASBL, Brussels
  - Hôpital Erasme,, Brussels
- Aarhus University Hospital, Aarhus N, Denmark
- Helsinki University Central Hospital, Helsinki, Finland
- Hospices Civils de Lyon, Hôpital Edouard Herriot, Lyon, France
- Germany (4):
  - Evangelisches Krankenhaus Düsseldorf, Düsseldorf
  - Universitätsklinikum Erlangen, Erlangen
  - Klinikum rechts der Isar, Münich
  - Sana Klinikum Offenbach GmbH, Offenbach
- OUS-Rikshospitalet University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Beyna T, Moreels T, Arvanitakis M, Pioche M, Saurin JC, May A, Knabe M, Agnholt JS, Bjerregaard NC, Puustinen L, Schlag C, Aabakken L, Paulsen V, Schneider M, Neurath MF, Rath T, Deviere J, Neuhaus H. Motorized spiral enteroscopy: results of an international multicenter prospective observational clinical study in patients with normal and altered gastrointestinal anatomy. Endoscopy. 2022 Dec;54(12):1147-1155. doi: 10.1055/a-1831-6215. Epub 2022 Apr 21. PMID 35451040

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm: Patients who received at least one procedure with the Motorized Spiral Endoscope (PowerSpiral).
Period: Overall Study
Arm/Group | Single Arm
Started | 302
Completed | 302
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 302 patient were enrolled, however 4 patients excluded because there was no deep enteroscopy conducted. So that 298 patients were analyzed according SAP.
Arm/Group | Single Arm
Number analyzed (Participants) | 298
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 122
  >=65 years | 176
Age, Continuous [Median (Full Range); unit: years] | 68 [19 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120
  Male | 178
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 298

OUTCOME MEASURES:

1. Primary Outcome: Collect Serious Adverse Events and Device Deficiencies to Demonstrate Safety of the Motorized Spiral Endoscope (PowerSpiral) in Daily Medical Practice.
Description: It is assumed that the new device and its safety profile is non-inferior to preceding generations of balloon assisted enteroscopes. Endoscope (PowerSpiral) in a typical clinical setting within the Intended Use
Time Frame: up to 12 days
Population: SAE rate
Measure: Number; unit: participants
Arm/Group | Single Arm
Number analyzed (Participants) | 298
participants
  Serious Adverse Events | 6
  Device Deficiencies | 1

2. Secondary Outcome: Number of Participants With Therapeutic Yield
Description: Defined as the percentage of patients with any endoscopic intervention / therapy with the exception of biopsies.
Time Frame: up to 12 days
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 298
Participants | 172

3. Secondary Outcome: Number of Participants With Procedures That Confirmed Previous Diagnosis
Description: Defined as the percentage of procedures that either confirmed a diagnosis from previous studies, or established a new definitive diagnosis at the anatomical location identified in previous studies or findings that could explain the clinical symptoms.
Time Frame: up to 12 days
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 298
Participants | 251

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the whole study duration of approx. 18 months and for each individual patients from signing the consent until hospital discharge.
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 7/298
Serious Adverse Events (participants affected / at risk) | 7/298
Other Adverse Events (participants affected / at risk) | 9/298
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=298)
Perforation (Gastrointestinal disorders) | 2 (2) — SAE occurred during the first procedure with PowerSpiral.
Bleeding (Gastrointestinal disorders) | 2 (2) — SAE occurred during the first and second procedure with PowerSpiral.
Mucosal injury (Gastrointestinal disorders) | 1 (1) — First procedure with PowerSpiral
Complications associated with sedation/anesthesia (General disorders) | 1 (1) — First and second procedure with PowerSpiral
Other (Gastrointestinal disorders) | 1 (1) — First procedure with PowerSpiral
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=298)
Bleeding (Gastrointestinal disorders) | 9 (9) — First procedure with PowerSpiral
Laceration (Gastrointestinal disorders) | 4 (4) — First and second procedure with PowerSpiral

LIMITATIONS AND CAVEATS:
Further evaluations of PowerSpiral in prospective studies in special indications like biliopancreatic interventions are needed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-04-23): https://cdn.clinicaltrials.gov/large-docs/81/NCT03955081/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-25): https://cdn.clinicaltrials.gov/large-docs/81/NCT03955081/SAP_001.pdf